CLINICAL TRIAL: NCT00059449
Title: Role of Epidermal Growth Factor (EGF) in Development of Necrotizing Enterocolitis
Status: Completed | Type: Observational
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Other Study IDs: EGFDNE (completed)
Record Dates: First submitted 2003-04-25; First posted 2003-04-29 (Estimated); Last update posted 2010-01-13 (Estimated); Status verified 2010-01

CONDITIONS: Necrotizing Enterocolitis; Premature Birth
Keywords: Enterocolitis
MeSH Terms: conditions — Enterocolitis, Necrotizing; Premature Birth; Enterocolitis

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Necrotizing enterocolitis (NEC) is a serious gastrointestinal disorder that primarily affects preterm infants. About 10% of babies less than 32 weeks gestation at birth will develop it. Overall, 30% of babies who develop NEC will die from it, with many others developing long term gastrointestinal problems. The most important factor in its development is a premature intestinal tract. Epidermal growth factor (EGF) is an important growth factor in the development and maintenance of the gastrointestinal tract. This study will look for a relationship between EGF levels in premature babies and the development of NEC.

ELIGIBILITY:
Inclusion Criteria:

* Gestational Age greater than 23 weeks at birth
* Birth weight greater than 500 grams
* Age less than 72 hours of life

Max Age: 72 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 372 (Estimated)

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Good Samaritan Hospital, Cincinnati, Ohio
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - University Hospital, Cincinnati, Ohio